

Name and surname:

Klinika Położnictwa, Perinatologii i Neonatologii CMKP

SPZOZ - Szpital Bielański im. ks. Jerzego Popiełuszki

01-809 Warszawa, ul. Cegłowska 80

tel. +48 (22) 56 - 90 - 274

Kierownik Kliniki: dr hab. n. med. Katarzyna Kosińska-Kaczyńska, prof. CMKP

28.02.2022

Comparison of the Efficacy of Emergency Two-level and Single Cervical Cerclage in Cervical Insufficiency in the Second Trimester of Pregnancy - Multicenter Prospective Randomized Trial

Cervical Occlusion Two-level Stitch Application (COSA)

Study Protocol and Statistical Analysis Plan Unique Protocol ID: nr 5/2024 7.04.2024

## DECLARATION OF CONSENT TO PARTICIPATE IN A MEDICAL EXPERIMENT

Head of the experiment: Dr hab. n. med. Katarzyna Kosińska-Kaczyńska, prof. CMKP

| 2. I was informed by | pation in the medical experiment is voluntary. withdraw my consent from this ] experiment at any time, ision will not result in any penalties or loss of any other prehensive and satisfactory answers to the questions I will have any questions or doubts during the experiment, or members of the research team. |
|---|---|
| or 1 resumently agree to postation | |
| <br>Date | Signature |